CLINICAL TRIAL: NCT06550336
Title: A Prospective, Single-center, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Chidamide Monotherapy for Maintenance Therapy in CD30+ Peripheral T-cell Lymphoma (PTCL).
Brief Title: A Clinical Study Assessing the Efficacy of Chidamide for CD30-positive Peripheral T-cell Lymphoma (PTCL).
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, Director, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: PTCL; chidamide
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: Chidamide tablets,the medication is to be taken at a dose of 20 mg (4 tablets) twice a week, specifically on days 1, 4, 8, 11, 15, 18, 22, and 25. It should be administered orally 30 minutes after meals.
  Treatment Duration: Each 4-week period constitutes one treatment cycle. Throughout the trial, all participants will continue to receive treatment until any of the following occurs: disease progression, intolerable adverse reactions, or the participant decides to withdraw.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide maintenance arm (Experimental): 20 mg (4 tablets) twice a week, specifically on days 1, 4, 8, 11, 15, 18, 22, and 25. It should be administered orally 30 minutes after meals.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — 20 mg (4 tablets) twice a week, specifically on days 1, 4, 8, 11, 15, 18, 22, and 25.Each 4-week period constitutes one treatment cycle.

SUMMARY:
* Objective:This study aims to assess the efficacy and safety of Chidamide as a monotherapy maintenance treatment for patients with newly diagnosed peripheral T-cell lymphoma (PTCL) who have achieved remission or stable disease after initial brentuximab vedotin (BV) plus cyclophosphamide, doxorubicin and prednisone (CHP)treatment, excluding ALK+ anaplastic large-cell lymphoma (ALCL).
* Design: The study is a prospective, single-center, open-label clinical trial.
* Treatment:Eligible patients will receive Chidamide tablets at a dosage of 20 mg (4 tablets) twice weekly. Treatment cycles are 4 weeks long and will continue until disease progression, unacceptable toxicity, patient withdrawal, investigator decision to discontinue, loss to follow-up, death, or study termination.
* Endpoints:The primary endpoint is the 2-year progression-free survival (PFS). Secondary endpoints include the overall response rate (ORR), overall survival (OS), and safety indicators.
* Rationale:The study seeks to provide a basis for the dosing regimen of Chidamide and contribute to the development of effective maintenance treatment strategies for PTCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. According to the WHO 2016 diagnostic criteria, the histological diagnosis is confirmed as CD30+ peripheral T-cell lymphoma (PTCL), including peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALK- ALCL), enteropathy-associated T-cell lymphoma (EATL), and other pathological subtypes (excluding extranodal NK/T-cell lymphoma, nasal type [NKTCL]). Patients with newly diagnosed PTCL (excluding ALK+ ALCL), who have completed 6 cycles of first-line treatment regimens (including various first-line induction chemotherapy regimens, targeted drugs, other treatment plans, and various combined therapies, etc.; with or without the inclusion of Chidamide) and have achieved complete remission (CR), and are not suitable for or do not consider undergoing autologous hematopoietic stem cell transplantation. Within 12 weeks from the first day of the last cycle of their first-line treatment regimen, they start to receive the medication plan of this study.
2. Age ≥18 years, male or female is not limited;
3. ECOG performance status score 0-3;
4. Neutrophils ≥1.5×10^9/L, platelets ≥80×10^9/L, hemoglobin ≥90g/L;
5. Expected survival time ≥3 months;
6. Voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women and women of childbearing age who are unwilling to adopt contraceptive measures;
2. Patients with a history of clinically significant prolongation of the QTc interval (males > 450ms, females > 470ms), ventricular tachycardia (VT), atrial fibrillation (AF), cardiac conduction block, myocardial infarction within the past year, congestive heart failure (CHF), and patients with symptomatic coronary artery disease requiring medication;
3. Patients who have undergone organ transplantation;
4. Patients who have received symptomatic treatment for previous bone marrow toxicity within 7 days prior to enrollment;
5. Patients with active bleeding;
6. Patients with a history of thrombosis, embolism, cerebral hemorrhage, cerebral infarction, or other related diseases;
7. Patients with active infection or those who have had persistent fever within 14 days prior to enrollment;
8. Patients who have undergone major organ surgery within the past 6 weeks;
9. Patients with abnormal liver function (total bilirubin > 1.5 times the normal value, ALT/AST > 2.5 times the normal value, or in liver-infiltrated patients ALT/AST > 5 times the normal value), and abnormal kidney function (serum creatinine > 1.5 times the normal value);
10. Patients with mental disorders/those who are unable to give informed consent;
11. Patients with drug abuse or chronic alcoholism that affects the evaluation of the trial results;
12. Patients with lymphoma involving the central nervous system;
13. Patients deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) rate | 24months
  PFS was defined as the time between diagnosis and the first date of relapse or all-cause death, whichever occurred first.

SECONDARY OUTCOMES:
overall survival (OS) | 48months
  OS was defined as the time after the date of diagnosis until all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No